CLINICAL TRIAL: NCT06225635
Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Ezerosu Tab. 10/20 mg(Single-layer Tablet) Compared to Ezerosu Tab. 10/20 mg(Double-layer Tablet) in Healthy Adult Volunteers
Brief Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Ezerosu Tab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP-RE-HYP-101
Record Dates: First submitted 2021-12-13; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2022-03

CONDITIONS: Hyperlipidemias
Keywords: Arteriosclerosis; Primary Hypercholesterolemia; Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias; Arteriosclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Ezerosu tablet(double layer tablet)
  Interventions: Drug: Ezerosu(monolayer tablet); Drug: Ezerosu(double layer tablet)
- Control (Active Comparator): Ezerosu tablet(monolayer tablet)
  Interventions: Drug: Ezerosu(monolayer tablet); Drug: Ezerosu(double layer tablet)

INTERVENTIONS:
Drug: Ezerosu(monolayer tablet) — Ezetimibe 10mg, Rosuvastatin calcium 20.8mg(20mg as Rosuvastatin)
Drug: Ezerosu(double layer tablet) — Ezetimibe 10mg, Rosuvastatin calcium 20.8mg(20mg as Rosuvastatin)

SUMMARY:
A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Ezerosu Tab

DETAILED DESCRIPTION:
Evaluate the Safety

1. Adverse Events
2. Concomitant Medications
3. Vital Signs
4. Laboratory Test

Pharmacokinetics

1. 1st Evaluation Variable: 1st Cmax, AUCt of Total Ezetimibe, Rosuvastatin
2. 2nd Evaluation Variable: AUC∞, Tmax, t1/2 of Total Ezetimibe, Rosuvastatin and Cmax, AUCt, AUC∞, Tmax, t1/2 of Free Ezetimibe

ELIGIBILITY:
Inclusion Criteria:

1. Those who are 19 years old or older at the time of the screening visit
2. At the time of screening visit, those who weigh 50 kg or more for men, 45 kg or more for women, and have a body mass index (BMI) of 18.0 kg / m2 or more and 30.0 kg / m2 or less.

   ☞ BMI (kg / m2) = Weight (kg) / {Height (m)} 2
3. Those who have no clinically significant congenital or chronic illness at the time of the screening visit and have no medical examination results, pathological symptoms or findings.
4. Diagnostic tests such as hematology tests, blood chemistry tests, serum tests, urine tests, and electrocardiogram test result tests set and performed by the test director (or the commissioned doctor in charge of the test) according to the characteristics of the clinical test drug. Now that it has been determined to fit the subject
5. Clinical trial drug From the first dosing date to the last clinical trial drug 14 days from the dosing date, the person, sperm, or partner should use medically appropriate contraceptive methods * to eliminate the possibility of pregnancy. Agree and agree not to donate sperm or eggs

   * Contraceptives: Combined use or killing of intrauterine devices, sperm surgery, tubal contraception and blockage contraceptives (male condoms, female condoms, cervical caps, contraceptive diaphragms, sponges, etc.) When using spermicide, use two or more contraceptive methods as a combination
6. A person who has signed a consent form by a free doctor after listening to and understanding the purpose and content of this clinical trial, the characteristics of the drug for clinical trial, expected abnormal reactions, etc.

Exclusion Criteria:

1. Digestive system, cardiovascular system, endocrine system, respiratory system, blood / tumor, infectious disease, kidney and urogenital system, psychiatric / nervous system, musculoskeletal system, immune system, otolaryngology, dermatology, ophthalmology People with clinically significant illness or past strength who fall into the system
2. Those who have past ability of gastrointestinal surgery (excluding simple appendectomy and hernia surgery) that can affect drug absorption, or have gastrointestinal illness
3. Those who took drug-metabolizing enzyme-inducing and inhibitory drugs such as barbital drugs within 1 month of the first dosing date, or took drugs that may interfere with this clinical study within 10 days of the first dosing date (however) , Interaction with clinical study drugs, half-life of concomitant drugs, etc. Can be participated in consideration of drug dynamics and pharmacodynamics)
4. Those who participated in other clinical trials or bioequivalence studies and received clinical trial drugs within 6 months of the first dosing date.
5. Those who donated whole blood or component blood within 2 weeks or received blood transfusion within 4 weeks on the first dosing day
6. Those who meet the following conditions within one month of the first dosing date

   * For men, alcohol intake exceeding 21 cups / week on average
   * For females, alcohol intake exceeding 14 cups / week on average

     (1 cup = 50 mL of shochu or 30 mL of Western liquor or 250 mL of beer)
   * Smoking an average of 20 cigarettes or more per day
7. Those who fall under the following

   ・ Persons with hypersensitivity to the main ingredients or constituents of this drug

   • Persons with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
8. Patients with the following diseases

   * Patients with active liver disease or patients with persistently high symptoms due to unknown causes of serum amino transduction enzyme levels
   * Patients with muscle disease
   * Patients receiving cyclosporine in combination
   * Patients with moderate renal disorder or severe renal failure (eGFR <60 ml / min / 1.73 m2)
   * Patients who are susceptible to myopathy and rhabdomyolysis
   * Patients with hypothyroidism
   * Patients with a history of genetic muscle disease or family history

     -Patients with a history of muscle toxicity to statins (HMG-CoA convertase inhibitors) or fibrates
   * Alcoholics
   * Patients treated with fibrates
9. Persons who are judged by the investigator (or the commissioned investigator) to be unsuitable for participation in this clinical study due to reasons other than the above selection / exclusion criteria.
10. In the case of female applicants, pregnant women or those who are suspected of becoming pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Cmax of Total Ezetimibe, Rosuvastatin | follow up to Day8
  Cmax of Total Ezetimibe, Rosuvastatin
AUCt of Total Ezetimibe, Rosuvastatin | follow up to Day8
  AUCt of Total Ezetimibe, Rosuvastatin

SECONDARY OUTCOMES:
AUC∞ of Total Ezetimibe, Rosuvastatin and AUC∞ of Free Ezetimibe | follow up to Day8
  AUC∞ of Total Ezetimibe, Rosuvastatin and AUC∞ of Free Ezetimibe
Tmax of Total Ezetimibe, Rosuvastatin and Tmax of Free Ezetimibe | follow up to Day8
  Tmax of Total Ezetimibe, Rosuvastatin and Tmax of Free Ezetimibe
t1/2 of Total Ezetimibe, Rosuvastatin and t1/2 of Free Ezetimibe | follow up to Day8
  t1/2 of Total Ezetimibe, Rosuvastatin and t1/2 of Free Ezetimibe
Cmax of Free Ezetimibe | follow up to Day8
  Cmax of Free Ezetimibe
AUCt of Free Ezetimibe | follow up to Day8
  AUCt of Free Ezetimibe

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea